CLINICAL TRIAL: NCT05980260
Title: Optimizing Pharmacologic Treatment for Neonatal Opioid Withdrawal Syndrome (OPTimize NOW): A Symptom-Based Dosing Approach
Acronym: OPTimize NOW
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: HELP for NOWS Consortium (Network)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HELP for NOWS 02; 1U24HD107621 (NIH); 1UG1HD107628 (NIH); 1UG1HD107580 (NIH); 1UG1HD107649 (NIH); 1UG1HD107650 (NIH); 1UG1HD107653 (NIH); 1UG1HD107627 (NIH); 1UG1HD107631 (NIH); 1UG1HD107616 (NIH)
Record Dates: First submitted 2023-07-27; First posted 2023-08-07 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Neonatal Opiate Withdrawal Syndrome
Keywords: NOWS

STUDY DESIGN:
Intervention Model Description: A two-period cluster crossover design will be used in this study. Study sites will be randomized in a 1:1 allocation ratio to one of two sequences:
  1. A three-week run-in period followed by a scheduled opioid taper approach for five months followed by a three-week washout period followed by a symptom-based dosing approach for five months.
  2. A three-week run-in period followed by a symptom-based dosing approach for five months followed by a three-week washout period followed by a scheduled opioid taper approach for five months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Other): This sequence will assign eligible participants to a three-week run-in period followed by a scheduled opioid taper approach for five months followed by a three-week washout period followed by symptom-based dosing approach for five months.
  Interventions: Other: Symptom-based Dosing Approach; Other: Scheduled Opioid Taper Approach
- Sequence 2 (Other): This sequence will assign eligible participants to a three-week run-in period followed by a symptom-based dosing approach for five months followed by a three-week washout period followed by scheduled opioid taper approach for five months.
  Interventions: Other: Symptom-based Dosing Approach; Other: Scheduled Opioid Taper Approach

INTERVENTIONS:
Other: Symptom-based Dosing Approach — During this approach to care, all enrolled infants with NOWS at the study site will be treated with the symptom-based dosing approach if they meet the withdrawal threshold for pharmacologic treatment. Participants may receive up to 3 doses of the study site's preferred opioid during a 24-hour period to treat signs of withdrawal once the threshold for pharmacologic intervention is met. If a 4th dose is required within a 24-hour period, the study site will transition to the scheduled opioid taper algorithm used at the study site to complete the infant's pharmacologic treatment.
Other: Scheduled Opioid Taper Approach — During this approach to care, all enrolled infants with NOWS at the study site will be treated with the study site's usual scheduled opioid taper approach, as detailed in each site's treatment algorithm, if they meet the withdrawal threshold for pharmacologic treatment.

SUMMARY:
This clinical trial will help us learn more about how to best care for babies with Neonatal Opioid Withdrawal Syndrome, also called NOWS. Babies with NOWS often have tremors, a hard time sleeping, excessive crying, and trouble feeding. Some babies that have NOWS need medicine. Doctors have two ways of providing medicine that are widely used today:

1. Scheduled opioid taper approach. The baby gets medicine at regular times. As symptoms get better, the amount of medicine the baby gets decreases until the baby no longer needs medicine. This is called a medicine taper.
2. Symptom-based approach. The baby will only get medicine when they show signs of NOWS, instead of at regular times. If the baby is showing no signs of NOWS, no medicine will be given.

We are doing the OPTimize NOW study to figure out the best way to give medicine to babies with NOWS.

DETAILED DESCRIPTION:
This two-period cluster crossover clinical trial will compare the length of time from birth until medically ready for discharge between infants with neonatal opioid withdrawal syndrome (NOWS) who are ≥ 36 weeks' gestation, at risk for pharmacologic treatment, and treated for NOWS with either a symptom-based dosing approach or a scheduled opioid taper approach.

Each study site (i.e., cluster) will be randomized in a 1:1 allocation ratio to one of two sequences:

* A three-week run-in period followed by a scheduled opioid taper approach for five months (Period 1) followed by a three-week washout period followed by a symptom-based dosing approach for five months (Period 2)
* A three-week run-in period followed by a symptom-based dosing approach for five months (Period 1) followed by a three-week washout period followed by scheduled opioid taper approach for five months (Period 2)

The randomization scheme will be stratified by the assessment and management approach used at each study site (i.e., Finnegan or Eat, Seep and Console).

ELIGIBILITY:
Inclusion Criteria:

1. The infant is greater than or equal to 36 weeks gestation.
2. The infant had antenatal opioid exposure identified by at least one of the following:

   * History of maternal opioid use during pregnancy;
   * Positive maternal toxicology screen for opioids during the second or third trimester of pregnancy; and/or
   * Positive infant toxicology screen for opioids during the initial hospital stay.
3. The infant is being assessed and managed for NOWS at an eligible study site.
4. The infant is at risk for pharmacologic treatment for NOWS defined by either of the following

   * At least 1 score ≥ 8 if assessed and managed with FNAST or modification thereof
   * At least 1 "yes" if assessed and managed with the ESC care approach

Exclusion Criteria:

1. The infant has major birth defect(s).
2. The infant has neonatal encephalopathy (inclusive of hypoxic ischemic encephalopathy), a metabolic disorder, stroke, intracranial hemorrhage, or meningitis diagnosed prior to the initiation of pharmacologic treatment.
3. The infant is receiving respiratory support (any positive pressure or oxygen therapy) at 48 hours of age.
4. The infant has undergone major surgical intervention prior to or at 48 hours of age.
5. The infant has postnatal opioid exposure prior to the initiation of treatment for NOWS.
6. The infant was outborn and pharmacologic treatment was initiated at the transferring hospital.
7. The infant is assessed for eligibility during the study site's three-week washout period.

Ages: 1 Hour to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-08-27 (Estimated)

PRIMARY OUTCOMES:
Time from birth until medically ready for discharge | From date of birth until hospital discharge or 1 year, whichever comes first.
  Time from birth until infant meets criteria for medically ready for discharge (days). An infant is considered medically ready for discharge when they are discharged by the medical provider or when they meet the following criteria the following criteria:
  * ≥ 96 hours of age
  * ≥ 48 hours since last dose of opioid treatment (i.e., morphine, methadone, or buprenorphine)

SECONDARY OUTCOMES:
Receipt of pharmacologic treatment | From date of birth until hospital discharge or 1 year, whichever comes first.
  If the infant received opioid replacement therapy prior to hospital discharge.
Length of hospital stay | From date of birth until hospital discharge or 1 year, whichever comes first.
  Number of days infant remained in the hospital
Safety outcomes | From date of birth until 3 months of life
  Safety outcomes including presence or absence of inpatient seizures, excessive weight loss of more than 15% from birthweight, and non-accidental trauma and death, and outpatient acute/urgent care or emergency room visits, hospital readmissions, and non-accidental trauma and death
Total number opioid doses | From date of birth until hospital discharge or 1 year, whichever comes first.
  The total number of opioid doses administered among all infants pharmacologically treated during initial hospitalization.
Receipt of secondary medications | From date of birth until hospital discharge or 1 year, whichever comes first.
  The total number of secondary opioid doses administered among all infants pharmacologically treated during intital hospitalization.
Transition from treatment with a symptom-based dosing approach to a scheduled opioid taper approach | From date of birth until hospital discharge or 1 year, whichever comes first.
  The total number of infants pharmacologically treated during intital hospitalization who transitioned from a symptom-based dosing approach to a scheduled opioid taper approach
Stopped scheduled opioid taper treatment | From date of birth until hospital discharge or 1 year, whichever comes first.
  The total number of infants pharmacologically treated during intital hospitalization who were initially treated with a scheduled opioid taper but stopped treatment due to excessive sedation or respiratory depression
Safety outcomes | From date of birth until hospital discharge or 1 year, whichever comes first.
  Safety outcomes among infants pharmacologically treated during initial hospitalization including presence or absence of inpatient seizures, excessive weight loss of more than 15% from birthweight, and non-accidental trauma and death, and outpatient acute/urgent care or emergency room visits, hospital readmissions, and non-accidental trauma and death

CONTACTS AND LOCATIONS:
Overall Officials: Lori Devlin, MD, Principal Investigator — University of Louisville
Locations (23):
- United States (23):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - ChristianaCare, Wilmington, Delaware
  - University of South Florida Health, Tampa, Florida
  - Sidney & Lois Eskenazi Hospital, Indianapolis, Indiana
  - University of Louisville Hospital, Jeffersonville, Indiana
  - University of Kansas Hospital, Kansas City, Kansas
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Kentucky Children's Hospital, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Norton Women's and Children's Hospital, Louisville, Kentucky
  - University of Nebraska Medical Center, Omaha, Nebraska
  - AtlantiCare Regional Medical Center, Atlantic City, New Jersey
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - University of Rochester Medical Center, Rochester, New York
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Kettering Health Main Campus, Kettering, Ohio
  - Oklahoma Children's Hospital OU Health, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Utah Health, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be analyzed and stored at the DCC, RTI International. NIH Helping to End Addiction Long-term Initiative (HEAL) and NICHD requirements for data-sharing will apply. NIH has had a long-standing policy to share and make available to the public the results and accomplishments of the activities that it funds. In accordance with these policies (available at HEAL Public Access and Data Sharing | NIH HEAL Initiative), we will share de-identified data collected for the study. After the study is completed, the de-identified, archived data will be transmitted to a NIH HEAL supported repository, for use by other researchers including those outside of the study.
Supporting Information: Study Protocol, SAP
Time Frame: Within 1 year of study completion.

REFERENCES:
- [Derived] Young LW, Babineau DC, Das A, DeMauro S, Kraft WK, Lorch S, Walsh MC, Merhar S, Devlin LA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research and the National Institutes of Health (NIH) Helping to End Addiction Long-term (HEAL) Initiative. Optimizing pharmacologic treatment for neonatal opioid withdrawal syndrome (OPTimize NOW): a symptom-based dosing approach study protocol for a multi-center, cluster crossover design randomized controlled trial. Trials. 2025 Aug 27;26(1):317. doi: 10.1186/s13063-025-09035-x. PMID 40866977
- See also: Related Info — http://helpfornows.rti.org